CLINICAL TRIAL: NCT03763422
Title: IDH Mutated 1p/19q Intact Lower Grade Glioma Following Resection: Wait Or Treat? IWOT - a Phase III Study
Brief Title: Trial in Low Grade Glioma Patients: Wait or Treat
Acronym: IWOT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poorly recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Cooperative Trials Group for Neuro-Oncology (COGNO) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-BTG-1635
Record Dates: First submitted 2018-11-13; First posted 2018-12-04 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Low-grade Glioma; Temozolomide; Phase III; Wait or Treat
MeSH Terms: interventions — Temozolomide; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Treatment arm (Experimental): Radiotherapy + Temozolomide
  Interventions: Drug: Temozolomide; Radiation: Radiotherapy
- Active surveillance arm (Active Comparator): Treatment as per local practice
  Interventions: Drug: Temozolomide; Radiation: Radiotherapy; Procedure: Surgery

INTERVENTIONS:
Drug: Temozolomide — Oral Administration of Temozolomide
  Other Names: TMZ
Radiation: Radiotherapy — 50.4 Gy in 28 fractions over 6 weeks
  Other Names: RT
Procedure: Surgery — Surgery
  Arms: Active surveillance arm

SUMMARY:
The 1635-EORTC-BTG study - Wait or Treat - concerns patients that represent a clinically favorable group of patients with IDHmutated astrocytoma (oligo-symptomatic), without a need for immediate post-operative treatment. It will establish whether early adjuvant treatment with radiotherapy and adjuvant temozolomide in resected IDHmutated astrocytoma will improve outcome, and whether benefits of early treatment outweigh potential side-effects of that, such as deterioration in neurocognitive function or Quality of Live, seizure activity and Patient Reported outcome compared to active surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Histologically WHO grade II (diffuse) or III (anaplastic) astrocytoma, IDHmt without 1p/19q co-deletion (local diagnosis)
* Time since diagnostic surgery or first resection ≤ 6 months
* No need for immediate radiotherapy followed by chemotherapy
* Having seizures only, without functional deficits due to the tumor (but the presence of functional deficits due to the resection is allowed)
* Patients for whom by local judgment an active surveillance policy is a realistic management alternative
* The patient is at least 18 years of age on day of signing informed consent
* WHO PS 0-2
* Adequate hematological, renal, and hepatic function, as follows:

  * Absolute neutrophil count ≥ 1.5 x 10*9/L
  * Platelets ≥ 100 × 10*9/L
  * Serum creatinine ≤ 1.5 times upper limit of laboratory normal (ULN)
  * Total serum bilirubin ≤ 1.5 × ULN
  * AST and ALT ≤ 2.5 × ULN
  * Alkaline phosphatase of ≤ 2.5 × ULN
* Presence of at least one paraffin block from the initial diagnosis for pathology review and translational research. If a representative formalin-fixed, paraffin-embedded (FFPE) block is not available, the collection of optimally 36, minimally 24 x 5 µm, unstained slides is required.
* At the time of randomization presence only of a non-enhancing tumor on T1 weighted contrast enhanced MR images; some faint non-nodular enhancement or enhancement that can be ascribed to the surgical resection or peri-operative ischemia is allowed. Preoperative enhancement is allowed provided this area is resected as shown on postoperative imaging
* Ability to take oral medication
* Women of child bearing potential (WOCBP) must have a negative serum or urine pregnancy test done within 72 hours prior to randomization
* Patients of childbearing / reproductive potential must agree to use adequate birth control measures, as defined by the investigator, during RT and TMZ treatment and for at least 6 months after the last TMZ cycle. A highly effective method of birth control is defined as those which result in low failure rate (i.e., less than 1 percent per year) when used consistently and correctly
* Women who are breast feeding must agree to discontinue nursing prior to the first dose of study treatment and until 6 months after the last study treatment
* Male patients should be advised not to father a child and not to donate sperm up to 6 months after receiving the last dose of TMZ, and to seek advice on cryoconservation of sperm prior to treatment start
* Ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and return for the required assessments
* Before patient registration/randomization, written informed consent must be given according to ICH/GCP, and national/local regulations

Exclusion Criteria:

* Presence of signs of increased intracranial pressure after surgery
* Requirement of steroids for control of tumor symptoms
* Presence of uncontrolled seizures after surgery, defined as having both:

  * persistent seizures interfering with everyday life activities AND
  * failed three lines of anti-epileptic drug regimen, including at least one combination regimen
* Presence of contra-indications for radiotherapy
* Hypersensitivity to dacarbazine (DTIC), to the active substance or to any of the excipients used for TMZ capsules
* Prior chemotherapy, or prior radiotherapy to the brain
* Pregnancy or breastfeeding
* Known HIV, chronic hepatitis B, or hepatitis C infection
* Inability to take oral medication (e.g., frequent vomiting, partial bowel obstruction)
* Concurrent severe or uncontrolled medical disease (e.g., active systemic infection, diabetes, hypertension, coronary artery disease, psychiatric disorder) that, in the opinion of the investigator, would compromise the safety of the patient or compromise the ability of the patient to complete the study
* Prior or second invasive malignancy, except non-melanoma skin cancer, completely resected cervical or prostate cancer (with PSA of less than or equal to 0.1 ng/mL). Other cancers for which the subject has completed potentially curative treatment more than 3 years prior to study entry are allowed
* Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2021-12-29 (Actual)

PRIMARY OUTCOMES:
Next intervention free survival (FIFS) | From the date of randomization until initiation of second treatment or death whichever occurs first assessed up to 11.5 years as of first patient in (FPI)

SECONDARY OUTCOMES:
First intervention free survival (FIFS) | from the date of randomization until initiation of preferably RT/TMZ or any other first therapeutic intervention (second surgery, RT, chemotherapy) or death (any cause) whichever occurs first assessed up to 11.5 years as of first patient in
Progression Free Survival (PFS) | From the date of randomization until the date of first objective progression or the date of patient's death whichever occurs first assessed up to 11.5 years as of first patient in
Overall Survival | From the date of randomization up to the date of death up to 1 year after first progression or start of second treatment in early treatment arm or first treatment in active surveillance arm assessed up to 11.5 years as of first patient in
Seizure activity | The IWOT Seizure Control Composite Score Index can be completed up to 4 weeks before or after the planned assessment. A time window of 8 weeks is therefore available for each assessment. Assessed up to 11.5 years after FPI
  Seizure activity will be evaluated by the IWOT Seizure Control Composite Score Index completed by patients with an additional answer from the local investigator.
Safety profile: CTCAE | The collection period will start from randomization and up to start of second treatment for patients in the early treatment arm and from randomization to first treatment, for patients in active surveillance arm. Assessed up to 11.5 years after FPI
  This study will use the International Common Terminology Criteria for Adverse Events (CTCAE), version 5.0, for adverse event reporting.
  Hematological toxicity will be assessed on the basis of blood counts. The nadir count will be assessed for each cycle of TMZ therapy, and graded according to CTCAE.
  Non-hematological acute side effects will be assessed and reported separately for each cycle of TMZ therapy, and graded according to the Common Terminology Criteria for Adverse Events version 5.0.
Translational research | tissue and blood at randomization and new tissue at repeated surgical interventions if patient consented for translational research.Assessed up to 11.5 years after FPI
  The main objectives of TR are the assessment of markers that can identify patients in whom an active surveillance policy is not recommended or who are at risk to develop delayed complications is important. Furthermore, identification of predictive factors that could guide when to start RT and chemotherapy would aid the implementation of an active surveillance approach in clinical practice.
HRQoL related to seizures | From randomization until progression assessed up to 11.5 years as of FPI
  A seizure specific questionnaire will be used. The Seizure Control Composite Score Index is self-reported 7-item questionnaire developed to assess seizures frequency and severity.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Van den Bent, Principal Investigator — EORTC Study Coordinator
Locations (45):
- Australia (10):
  - Princess Alexandra Hospital - University of Queensland, Woolloongabba, Brisbane, QLD
  - Prince of Wales Hospital, Randwick - Sydney, New South Wales
  - Westmead Hospital - Crown Princess Mary Cancer Centre, Westmead, New South Wales
  - Illawarra Cancer Care Centre - Wollongong Hospital, Wollongong, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Monash Medical Centre, Clayton, Victoria
  - St Vincent's Hospital, Fitzroy (Melbourne), Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Universitaetskliniken der Uni Wien - Universitaetsklinikum Wien - AKH uniklinieken, Vienna, Austria
- Belgium (2):
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - Gasthuiszusters van Antwerpen - GasthuisZusters Antwerpen - Sint-Augustinus, Wilrijk
- Aarhus University Hospitals - Aarhus University Hospital-Skejby, Aarhus, Denmark
- France (5):
  - CHU de Lyon - CHU Lyon - Hopital neurologique Pierre Wertheimer, Bron
  - CHRU de Lille, Lille
  - Assistance Publique - Hopitaux de Marseille - Hôpital de La Timone (APHM), Marseille
  - Assistance Publique - Hopitaux de Paris - La Pitie Salpetriere, Paris
  - Institut de Cancerologie Strasbourg Europe (formar Paul Strauss), Strasbourg
- Italy (7):
  - AUSL Bologna - Ospedale Bellaria, Bologna
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Istituto Clinico Humanitas, Milan
  - IRCCS - Istituto Neurologico Carlo Besta, Milan
  - IRCCS - Istituto Oncologico Veneto, Padua
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino - Ospedale San Giovanni - Dipartimento Neuroscienze, Torino
- Netherlands (7):
  - Catharina Ziekenhuis, Eindhoven
  - Leiden University Medical Centre, Leiden
  - Haaglanden Medisch Centrum (HMC) - Haaglanden MC - locatie Antoniushove, Leidschendam
  - Maastro Clinic - Maastricht Radiation Oncology, Maastricht
  - Erasmus MC, Rotterdam
  - ETZ Tilburg - St. Elisabethziekenhuis TweeSteden, Tilburg
  - UMC-Academisch Ziekenhuis Utrecht, Utrecht
- Spain (6):
  - Hospital Clinic Universitari de Barcelona, Barcelona
  - Institut Catala d'Oncologia - ICO L'Hospitalet - Hospital Duran i Reynals, Barcelona
  - Institut Catala d'Oncologia - Hospital Germans Trias i Pujol, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 De Octubre, Madrid
  - Hospital Universitario La Fe, Valencia
- Switzerland (3):
  - Oncology Institute of Southern Switzerland (IOSI), Bellinzona
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - UniversitaetsSpital Zurich, Zurich
- United Kingdom (3):
  - NHS Tayside - Ninewells Hospital, Dundee, Scotland
  - NHS Lothian - Western General Hospital, Edinburgh
  - Clatterbridge Centre for Oncology NHS Trust - Clatterbridge NHS -Wirral, Metropolitan Borough of Wirral